CLINICAL TRIAL: NCT06903117
Title: Clinical Study of CEA Targeting Chimeric Antigen Receptor T Lymphocytes (CAR-T) for CEA Positive Advanced Lung Cancer
Brief Title: Anti-CEA CAR-T for Advanced CEA-Positive Lung Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBC087
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Advanced Lung Cancer
Keywords: CEA; CAR-T

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Targeted CEA CAR-T intravenous infusion group (Experimental)
  Interventions: Biological: Targeted CEA CAR-T
- Targeting CEA CAR-T pleural infusion group (Experimental)
  Interventions: Biological: Targeted CEA CAR-T

INTERVENTIONS:
Biological: Targeted CEA CAR-T — Subjects meeting the transfusion criteria will receive pre-treatment, which is as follows: fludarabine 25mg/m2/d×3day and cyclophosphamide 300mg/m2/d×3day, and intravenous CEA CAR-T therapy after 1-2 days of rest
  Arms: Targeted CEA CAR-T intravenous infusion group
Biological: Targeted CEA CAR-T — Subjects meeting the reinfusion criteria will receive pre-treatment with fludarabine 25mg/m2/d×3day and cyclophosphamide 300mg/m2/d×3day, rest for 1-2 days, and intraperitoneal reinfusion targeted CEA CAR-T therapy
  Arms: Targeting CEA CAR-T pleural infusion group

SUMMARY:
Lung cancer is the leading cause of morbidity and mortality in the world, of which 80%-85% are non-small cell lung cancer (NSCLC). Most patients with NSCLC are at the advanced stage of diagnosis and have a poor prognosis. The 5-year survival rate of stage III patients is about 15%, the 5-year survival rate of stage IV patients is less than 5%, and the median survival time is only 7 months.

CEACAM5 (CEA), also known as CD66e, is a classic tumor marker that has been used as a marker for many types of tumors for 50 years. It is mainly expressed in lung cancer, esophageal cancer, bile duct cancer, colorectal cancer, gastric cancer and other tumor types.

In previous CAR-T-related clinical trials targeting CEA, the research team found that CAR-T cell preparations had a certain killing effect on CEA positive tumor cells. At the same time, CAR-T cell preparations cannot be sustained for a long time in the body, which is also a key factor restricting the anti-tumor effect of CAR-T cells in the body. To solve this problem, the killing ability and survival ability of CAR-T cell preparations on tumor cells in vitro and in vivo were improved by optimizing CAR structure and improving culture mode.

DETAILED DESCRIPTION:
This study is a single-arm, open, enhanced 3+3 dose-ascending + dose-extending clinical study, aiming to evaluate the safety and efficacy of CAR T cell preparations, initially observe and study the pharmacokinetic characteristics of drugs in CEA positive advanced lung cancer patients, and obtain the recommended dose of CAR T cell preparations for CEA positive advanced lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, male or female;
2. histologically or pathologically confirmed advanced, metastatic or recurrent lung cancer, including non-small cell lung cancer and small cell lung cancer;
3. Progression or intolerance (including but not limited to surgery, chemotherapy, radiotherapy, targeted therapy, immunotherapy, etc.) after receiving at least second-line standard therapy, patients with driver gene positive non-small cell lung cancer need to receive corresponding targeted therapy for disease progression or intolerance. Patients with driver negative non-small cell lung cancer or small cell lung cancer need to receive platinum-containing chemotherapy for disease progression or intolerance;
4. Immunohistochemical staining of tumor samples within 3 months confirmed CEA positive (clear membrane staining, positive rate ≥10%); If the immunohistochemical results of tumor samples are more than 3 months from the time of screening (clear membrane staining, positive rate ≥10%), the patient's serum CEA should exceed 10ug/L.
5. There is at least one evaluable lesion according to RECIST 1.1 criteria, and the length of the extranodal lesion should be ≥10mm; For nodular lesions, the short diameter of the lymph node should be ≥15mm.
6. ECOG score 0-2 points ;
7. The expected survival time is more than 12 weeks;
8. no serious mental disorders;
9. Unless otherwise stated, the subject's vital organ functions shall meet the following conditions:

   1. Blood routine: Neutrophils>1.0×109/L, platelet>75×109/L, hemoglobin > 80g/L;
   2. Cardiac function: Echocardiography indicated cardiac ejection fraction ≥50%, and no obvious abnormality was found in electrocardiogram;
   3. Renal function: serum creatinine ≤2.0×ULN;
   4. Liver function: ALT and AST≤3.0×ULN (patients with liver tumor infiltration can be relaxed to ≤5.0×ULN);
   5. Total bilirubin ≤2.0×ULN;
   6. Blood oxygen saturation in non-oxygen state>92%.
10. Have the criteria for simple or intravenous blood collection, and no other contraindications for cell collection;
11. The subject agrees to use a reliable and effective contraceptive method for contraception (excluding safe period contraception) for 1 year from signing the informed consent to receiving the CAR T cell infusion;
12. The patient or his/her guardian agrees to participate in the clinical trial and signs the ICF, indicating that he/she understands the purpose and procedure of the clinical trial and is willing to participate in the study.

Exclusion Criteria:

1. Patients with central nervous system metastasis or meningeal metastasis with clinical symptoms at the time of screening, or with other evidence that the central nervous system metastasis or meningeal metastasis was not controlled, and the investigators judged that they were not suitable for inclusion;
2. Participating in other clinical studies within 1 month before screening;
3. Received live attenuated vaccine within 4 weeks prior to screening;
4. have received any of the following anti-tumor therapies prior to screening: chemotherapy, targeted therapy, or other investigational agents within 14 days or at least 5 half-lives, whichever is shorter;
5. There is an active infection or uncontrollable infection that requires systemic treatment;
6. The tumor compresses the trachea or important large blood vessels, and the risk is greater as assessed by researchers;
7. There is a large number of uncontrollable fluid accumulation in the serous cavity;
8. Toxicity of previous antitumor therapy has not improved to baseline level or ≤ grade 1, except for alopecia or peripheral neuropathy;
9. Have any of the following heart conditions:

   1. New York Heart Association (NYHA) Stage III or IV congestive heart failure;
   2. Had myocardial infarction or coronary artery bypass grafting (CABG) within ≤6 months before enrollment;
   3. A history of clinically significant ventricular arrhythmia, or unexplained syncope (other than those caused by vasovagal or dehydration);
   4. History of severe non-ischemic cardiomyopathy;
10. Patients with active autoimmune diseases, or other patients requiring long-term immunosuppressive therapy;
11. Other uncured malignant tumors within the past 3 years or at the same time, except cervical carcinoma in situ and skin basal cell carcinoma;
12. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer greater than the normal range; Hepatitis C virus (HCV) antibody positive and peripheral blood hepatitis C virus (HCV) RNA detection greater than the normal range; Positive for human immunodeficiency virus (HIV) antibodies; Syphilis positive;
13. Women who are pregnant or breastfeeding;
14. Circumstances deemed unsuitable for participation in the study by other researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of CAR T cell preparations in the treatment of CEA positive advanced lung cancer【safety】 | 28days
  Adverse events and their proportion during the trial (assessed against the Common Terminology Standard for Adverse Events Version 5.0 (CTCAE 5.0) and ASTCT standards)

SECONDARY OUTCOMES:
To evaluate the disease control rate and remission rate of CAR-T cell preparations in CEA positive advanced lung cancer【efficacy】 | 3months
  1）Disease control rates at 3 months were assessed according to Response Evaluation Criteria in Solid Tumors,Version 1.1 (RECIST 1.1), including CR, PR, and SD； 2）Objective response rates at 3 months were assessed according to RECIST 1.1, including CR, PR；
To evaluate the survival benefit of CAR-T cell preparations in CEA-positive advanced lung cancer【efficacy】 | 2years
  1）Overall survival (OS) : The time from the time the subject received CAR T cell retransfusion until death (from any cause)； 2）Duration of response (DOR) : the time from the first evaluation of CR, PR, or SD to the first evaluation of disease recurrence or progression or death from any cause; 3）Disease progression-free survival (PFS) : the time from the time the subject received CAR T cell therapy until the first disease progression or death from any cause;
To obtain the cytodynamics data of CAR-T cells in vivo【pharmacokinetics】 | 3months
  Cmax:The highest concentration of CAR T cells amplified in peripheral blood after reinfusion
To obtain the cytodynamics data of CAR-T cells in vivo【pharmacokinetics】 | 3months
  Tmax:The time to reach the highest concentration of CAR-T cells in peripheral blood after reinfusion
To obtain the cytodynamics data of CAR-T cells in vivo【pharmacodynamics】 | 2years
  The content of free CEA in peripheral blood at each time point after transfusion was determined by immunohistochemical method

CONTACTS AND LOCATIONS:
Locations (1):
- Changzheng Hospital, Naval Military Medical University, Shanghai, China, Shanghai, China

IPD SHARING:
Plan to Share IPD: No